CLINICAL TRIAL: NCT00642304
Title: A Single Arm Open Label Study to Assess Efficacy, Safety and Tolerability of Once-monthly Administration of Subcutaneously C.E.R.A. for the Maintenance of Hemoglobin Levels in Patients With Chronic Renal Anemia Not on Dialysis
Brief Title: A Study of Subcutaneous C.E.R.A. for the Maintenance of Hemoglobin Levels in Participants With Chronic Renal Anemia Not on Dialysis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20937
Record Dates: First submitted 2008-03-19; First posted 2008-03-25 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- methoxy polyethylene glycol-epoetin beta (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [C.E.R.A.]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [C.E.R.A.] — Methoxy polyethylene glycol-epoetin beta is administered SC every four week up to Week 20.The starting dose is 120, 200 or 300 mcg based on the dose of darbepoetin alfa or epoetin beta participants shall be receiving in the week preceding the study start. Further dose adjustment during the study depending on the hemoglobin (Hb) values.

SUMMARY:
This single arm study will assess the efficacy and safety of subcutaneous C.E.R.A. when administered for the maintenance of hemoglobin levels in participants with chronic renal anemia, not on dialysis. Participants currently receiving maintenance treatment with subcutaneous darbepoetin alfa or epoetin beta will receive monthly injections of C.E.R.A., with the starting dose (120, 200 or 300 micrograms [mcg] subcutaneously [SC]) derived from the dose of darbepoetin alfa or epoetin beta they were receiving in the week preceding study start.

ELIGIBILITY:
Inclusion Criteria:

* Chronic renal anemia
* Stable darbepoetin alfa or epoetin beta therapy for past 8 weeks

Exclusion Criteria:

* Transfusion of red blood cells during previous 8 weeks
* Poorly controlled hypertension requiring interruption of epoetin treatment in previous 6 months
* Acute or chronic bleeding requiring therapy within previous 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-03-27 (Actual); Primary Completion 2009-12-09 (Actual); Study Completion 2009-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- Netherlands (23):
  - Twenteborg Ziekenhuis, Almelo
  - Meander Mc, Locatie Lichtenberg; Dept of Lung Diseases, Amersfoort
  - Bovenij Zkhs; Cardiologie Afd., Amsterdam
  - Wilhelmina Ziekenhuis; Inwendige Geneeskunde, Assen
  - Rode Kruis Ziekenhuis; Inwendige Geneeskunde, Beverwijk
  - Amphia Ziekenhuis, Breda
  - Reinier De Graaf Groep, Delft
  - Slingeland Ziekenhuis; Inwendige Geneeskunde, Doetinchem
  - Albert Schweitzer Ziekenhuis; Inwendige Geneeskunde, Dordrecht
  - Nij Smellinghe Ziekenhuis; Inwendige Geneeskunde, Drachten
  - Oosterscheldeziekenhuis, Goes
  - Groene Hart Ziekenhuis Bleulandlocatie; Inwendige Geneeskunde, Gouda
  - Atrium Medisch Centrum; Nephrology, Heerlen
  - Bethesda Hospital; Internal Medicine, Hoogeveen
  - Leiden University Medical Center; Nierziekten, Leiden
  - Rijnland Zkhs Loc Leiderdorp; Interne geneeskunde, Leiderdorp
  - Academish Ziekenhuis Maastricht (Azm); Inwendige Geneeskunde, Maastricht
  - Academisch Ziekenhuis St. Radboud; Nierziekten Afd., Nijmegen
  - Erasmus Mc - Locatie Centrum; Inwendige Geneeskunde, Rotterdam
  - Mc Rijnmond Zuid - Locatie Clara; Infectieziekten, Rotterdam
  - Ikazia Ziekenhuis; Interne Oncologie, Rotterdam
  - Zorgsaam Ziekenhuis, Terneuzen
  - Diakonessenhuis, Utrecht

RESULTS

PARTICIPANT FLOW:
Groups:
- Methoxy Polyethylene Glycol-epoetin Beta: Methoxy polyethylene glycol-epoetin beta was administered subcutaneously (SC) every four weeks up to Week 20. The starting dose was 120, 200 or 300 micrograms (mcg) based on the dose of darbepoetin alfa or epoetin beta they were receiving in the week preceding the study start. Further dose was adjusted during the study depending on the hemoglobin (Hb) levels.
Period: Overall Study
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Started | 20
Completed | 14
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Blood transfusion | 2
Not completed — Erythropoiesis Stimulating Agent Use. | 1
Not completed — Transplantation | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose trial medication and underwent a safety follow-up, whether withdrawn prematurely or not.
Groups:
- Methoxy Polyethylene Glycol-epoetin Beta: Methoxy polyethylene glycol-epoetin beta was administered SC every four weeks up to Week 20. The starting dose was 120, 200 or 300 mcg based on the dose of darbepoetin alfa or epoetin beta they were receiving in the week preceding the study start. Further dose was adjusted during the study depending on the Hb levels.
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (16.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Hb Concentration Within +/-1 Gram Per Deciliter (g/dL) of Their Reference Hb and Between 10.5 to 12.5 g/dL Throughout the Efficacy Evaluation Period (EEP)
Description: The reference Hb value was taken as the time adjusted average of all Hb assessments during the Stability Verification Period (SVP) (Week -4 to Week 0). EEP was from Week 16 to Week 24.
Time Frame: EEP (Weeks 16 to 24)
Population: The Intent- to -treat (ITT) population included all participants who received at least one dose of trial medication at Week 0 and for whom data for at least one follow-up variable (adverse event) was available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 20
Percentage of participants | 40 [19.1 to 64.0]

2. Secondary Outcome: Mean Change in Hb Concentration Between SVP and the EEP
Description: The mean change in the time-adjusted average Hb concentration between the two study periods SVP (Baseline) and EEP is presented. The SVP was defined as Week -4 to Week 0. The EEP was defined as Week 16 to Week 24.
Time Frame: SVP (Week -4 to Week 0) and EEP (Week 16 to Week 24)
Population: ITT population
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 20
g/dL | 0.2 (1.15)

3. Secondary Outcome: Percentage of Participants Maintaining Hb Concentration Within Hb Range 10.5 to 12.5 g/dL During the EEP
Description: The EEP was defined as Week 16 to Week 24.
Time Frame: EEP (Weeks 16 to 24)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 20
Percentage of participants | 50.0 [27.2 to 72.8]

4. Secondary Outcome: Mean Time Spent in Hb Range of 10.5 to 12.5 g/dL During the EEP
Description: The EEP was defined as Week 16 to Week 24.
Time Frame: EEP (Weeks 16 to 24)
Population: ITT population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 20
Days | 36.5 (24.4)

5. Secondary Outcome: Percentage of Participants With Blood Transfusion
Time Frame: Baseline up to Week 28
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 20
Percentage of participants | 10

6. Secondary Outcome: Percentage of Participants With Dose Adjustment
Description: A dose adjustment was defined as a change versus the preceding dose. It included dose increase and dose reduction from the dose given at Baseline.
Time Frame: Baseline up to Week 20
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Number analyzed (Participants) | 20
Percentage of participants | 60

ADVERSE EVENTS:
Time Frame: Baseline up to Week 28
Arm/Group | Methoxy Polyethylene Glycol-epoetin Beta
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (N=20)
Myocardial infarction (Cardiac disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 2
Blood Potassium increased (Investigations) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemodialysis (Surgical and medical procedures) | 1
Renal transplant (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-epoetin Beta (N=20)
Anaemia (Blood and lymphatic system disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Regurgitation (Gastrointestinal disorders) | 1
Hypothermia (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Erysipelas (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Blood calcium increased (Investigations) | 1
Blood phosphorus increased (Investigations) | 2
Blood potassium increased (Investigations) | 2
Blood pressure increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 2
Urinary bladder haemorrhage (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.